CLINICAL TRIAL: NCT02560714
Title: SI Joint Fusion and Decortication Using the SImmetry System
Status: Terminated | Type: Observational
Why Stopped: No additional enrollment
Sponsor: Zyga Technology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1099
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: sacroiliac joint fusion; SIJ Fusion; SI Joint; SIJ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SImmetry Sacroiliac Fusion System — SImmetry
  The SImmetry device is commercially available. The implanted devices consist of a range of threaded, self-tapping, cannulated implants designed to transfix the sacrum and ilium, providing stability for intra-articular fusion.
  The SImmetry Surgical Instruments include standard manual surgical instruments used to access and prepare the sacroiliac joint space for intra-articular fusion.

SUMMARY:
The purpose of the SI Joint Fusion and Decortication Using the SImmetry System study is to evaluate the SImmetry Sacroiliac Joint Fusion System for fusion of the SI joint and relief of SI joint pain symptoms.

DETAILED DESCRIPTION:
This is a prospective, non-randomized post market study designed to collect data on SI joint fusion and subject back pain following implant of the SImmetry device. The study will be conducted at a single site and 25 subjects will be implanted and followed through 24 months. Data will be collected pre-operatively, implant, and at specified follow-up time points through 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be indicated for the SImmetry device according to the approved SImmetry labeling
* Subject has two (2) positive (experiences pain) Provocative Tests for SIJ pain; for example, Compression, Thigh Thrust, FABER, Distraction or Gaenslen's
* Subject has documentation of failed, non-operative management of SIJ pain for ≥ 6 months prior to surgery; for example, use of medications, braces, SI belts, orthotics, physical therapy or manual manipulation
* The subject has two (2) diagnostic SIJ injection at least one (1) resulting in a ≥50% decrease in pain in the joint(s) from the anesthetic portion of the injection
* The subject has VAS back pain score of ≥ 50 mm
* The subject is at least 18 years of age and skeletally mature
* The subject agrees and is able to comply with study requirements

Exclusion Criteria:

* Subjects contraindicated per the cleared labeling will be excluded from participation in the study
* The subject has pelvic soft tissue or bony tumors
* The subject has had any trauma causing fracture of the sacrum or iliac bones or has had spinal trauma leading to a neurological deficit
* The subject has a history of a central nervous system (CNS) disorder(s)
* The subject is indicated for or awaiting other spine surgery
* The subject is pregnant or is planning on becoming pregnant in the next two years
* The subject has uncontrolled insulin dependent diabetes mellitus (Type 1 Diabetes)
* The subject has chemical dependency abuse problems as evidenced by a history of abusing drugs which is documented in their past medical history or is elicited from an interview
* The subject is receiving or seeking worker's compensation, disability remuneration, and/or involved in litigation related to low back or SIJ pain
* The subject has a history of significant emotional or psychosocial disturbance (untreated or uncontrolled anxiety attacks, obsessive/compulsive disorders, depression or schizophrenia) as documented in their past medical history or elicited by an interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Investigator's standard patient population diagnosed with SIJ pain and candidates for SIJ fusion.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
SI Joint Fusion | 24 months
  Number of participants with radiographic evidence of fusion of the SI joint, defined as presence of a continuous segment of solid bridging bone that extends from the sacrum to the ilium.
SI Joint Pain Reduction | 6 months
  SI joint pain reduction evaluated by use of Visual Analogue Scale (VAS) for back pain for comparison of baseline to 6 months.

SECONDARY OUTCOMES:
SI Joint Pain Reduction | 24 Months
  SI joint pain reduction evaluated by use of Visual Analogue Scale (VAS) for back pain for comparison of baseline to all follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Reno Orthaepedic Clinic, Reno, Nevada, United States